CLINICAL TRIAL: NCT06034418
Title: The Efficacy of Pulse Radiofrequency Treatment to Articular Branches of Femoral and Obturator Nerves in Patients With Coxarthrosis
Brief Title: Efficacy of Pulse Radiofrequency Treatment in Patients With Coxarthrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Fatıma Korkmaz, MD, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraCHBilkent-FTR-FK-01
Record Dates: First submitted 2023-08-22; First posted 2023-09-13 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Coxarthrosis; Primary
Keywords: coxarthrosis; pain; pulse radiofrequency; nerve block
MeSH Terms: conditions — Osteoarthritis, Hip; Pain | interventions — Nerve Block; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulse Radiofrequency Group (Active Comparator): Pulse radiofrequency therapy will be applied to each nerve in 2 cycles of 120 seconds for patients in the pulse radiofrequency group. After the pulse radiofrequency procedure, 1 cc betamethasone and 1 cc 1% lidocaine will be injected for each nerve.
  Interventions: Device: Pulse radiofrequency treatment; Drug: Nerve block with 1 cc betamethasone and 1 cc 1% lidocaine
- Block Group (Active Comparator): For the patients in the block group, nerve block will be performed by applying 1 cc betamethasone and 1 cc 1% lidocaine for each nerve.
  Interventions: Drug: Nerve block with 1 cc betamethasone and 1 cc 1% lidocaine

INTERVENTIONS:
Device: Pulse radiofrequency treatment — In the procedures to be performed under fluoroscopy, vascular structures will be detected primarily by ultrasonography for safety purposes. A standard RF device will be used for the process. A 22-gauge and 10 cm straight radiofrequency cannula with 1 cm active tip will be used. For each nerve, sensory stimulation will be performed at 50 Hz and the patient will be expected to feel numbness and tingling with a maximum 0.7 V. Motor stimulation will be at 2 Hz and no muscle contraction up to 2 V is expected. Following the appropriate cannula placement, pulse radiofrequency will be applied to each nerve in 2 cycles of 120 seconds for the patients in this group. The pulse radiofrequency current will be 20 milliseconds wide and 45 volts in size. The tip temperature shall not be more than 42℃.
  Arms: Pulse Radiofrequency Group
Drug: Nerve block with 1 cc betamethasone and 1 cc 1% lidocaine — In the procedures to be performed under fluoroscopy, vascular structures will be detected primarily by ultrasonography for safety purposes. A standard RF device will be used for the process. A 22-gauge and 10 cm straight radiofrequency cannula with 1 cm active tip will be used. For each nerve, sensory stimulation will be performed at 50 Hz and the patient will be expected to feel numbness and tingling with a maximum 0.7 V. Motor stimulation will be at 2 Hz and no muscle contraction up to 2 V is expected. Following the appropriate cannula placement, patients will be injected with 1 cc betamethasone and 1 cc 1% lidocaine for each nerve. A total of 2 cc volume will be injected for each nerve.

SUMMARY:
Our aim in this interventional study is to investigate the effectiveness of pulsed radiofrequency (PRF) treatment applied to the articular branches of the femoral and obturator nerves on pain, functional level, functional capacity and quality of life in patients with coxarthrosis. We will compare the effects of PRF treatment added to nerve block compared to nerve block alone.

DETAILED DESCRIPTION:
Hip pain caused by coxarthrosis is common in the general population and is one of the leading causes of disability in the aging population. Conservative treatments may fail due to side effects or ineffectiveness. Surgery is generally recommended for patients who do not respond to conservative treatment. Surgery is not always an appropriate option for elderly patients and patients with multiple comorbidities. For this reason, nerve block may be an appropriate treatment option for patients who do not respond to conservative treatment, who are not suitable for surgery or who do not want surgery. Pulsed radiofrequency (PRF) is a method of temporarily preventing pain transmission through heat increase in the tissue with the help of an electrode placed near the target nerve. Most of the pain sensation in the hip joint is received by the articular branches of the femoral and obturator nerves. The application of PRF to the nerves innervating the hip joint may be an effective method to reduce pain and disability in these patients.

This study was designed as a prospective, randomized, controlled trial. According to the statistical analysis, 28 patients who met the eligibility criteria were planned to be included in the study. The patients will be divided into 2 groups as the block group (n=14) and the PRF group (n=14). In procedures performed under fluoroscopy, vascular structures will be detected primarily by ultrasonography for safety purposes. Nerve block and PRF procedures will be performed in sterile conditions according to their protocols. Patients will be evaluated about pain, functional level, functional capacity and quality of life before treatment, at week 2, week 4, and week 12. If complications develop, they will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral and/or bilateral hip pain for more than 6 months who meet the diagnosis of coxarthrosis according to the American College of Rheumatology(ACR) criteria
* Pain intensity greater than 3 according to the visual analog pain scale
* Stage ≥2 hip osteoarthritis according to the Kellgren-Lawrence classification
* Ambulation with or without support
* Having the mental competence to express pain scores
* Signing an informed consent form stating consent to participate in the study

Exclusion Criteria:

* Other non-degenerative causes of hip pain (Avascular necrosis, femoraacetebular impingement syndrome, thoracenteric bursitis)
* Concomitant central nervous system and/or peripheral nervous system disease
* History of lower extremity fracture/surgery in the last 6 months
* Local infection on the hip or presence of systemic infection
* Conditions where fluoroscopy-guided injection is contraindicated like pregnancy, contrast material allergy, local anesthetic allergy, coagulopathy
* Presence of unstable systemic diseases

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | baseline, week 2, week 4 and week 12
  Visual Analogue Scale (VAS) is one of the pain rating scales. The amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain. The VAS consists of a 10 cm line, with two end points representing 0 (no pain) and 10 (extreme pain). At rest, with movement, nighttime VAS scores and averages of them will be recorded.

SECONDARY OUTCOMES:
Active Range of Motion | baseline, week 2, week 4 and week 12
  Active ROM is a joint movement that can be achieved by active muscle contraction without the aid of external forces. It will be measured with a goniometer by physician.
Passive Range of Motion | baseline, week 2, week 4 and week 12
  Passive ROM is joint motion that can be achieved with the help of external forces. It will be measured with a goniometer by physician.
Harris Hip Score (HHS) | baseline, week 2, week 4 and week 12
  HHS is a measure of dysfunction for the hip joint. It consists of 4 parts including pain, function, absence of deformity and range of motion. Scores range from 0 to 100. Higher scores mean less dysfunction.
Six Minute Walk Test | baseline, week 2, week 4 and week 12
  6-minute walk test is used to measure the functional capacity of the person. A 30-meter-long, flat and hard-floored walking path is used. The start and end points are marked with cones. The distance that walked over 6 minutes will be recorded. Higher distance indicates better functional capacity.
Short From-36 (SF-36) | baseline, week 2, week 4 and week 12
  Sf-36 is a questionare that measure health related quality of life. It includes 36 questions and assesses 8 health domains: physical functionality, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain and general health perceptions. Scores for each domain range from 0 to 100. A higher score identifies a better state of health.
Number of analgesics | baseline, week 2, week 4 and week 12
  The number of analgesic drugs used daily by the patient is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No